CLINICAL TRIAL: NCT02123251
Title: A Randomized Incentive-Based Diabetes Self-Management Study (Hawaii Patient Reward And Incentives to Support Empowerment Project)
Brief Title: Hawaii Patient Reward And Incentives to Support Empowerment
Acronym: HI-PRAISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); Hawaii Department of Human Services (DHS) (Unknown); Kaiser Permanente (Other); RTI International (Other); IMPAQ International, LLC. (Industry); Econometrica, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Rude Ozaki, Associate Professor, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDFA93.536 -CMS-MIPCD-HI; 1B1CMS330884-01 (Other Grant/Funding Number: CMS)
Record Dates: First submitted 2014-04-15; First posted 2014-04-25 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Incentives,; Diabetes,; Medicaid,; Health behavior,; Cost effectiveness
MeSH Terms: conditions — Diabetes Mellitus; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial Incentives Group (Experimental): Participants (159) in the Incentive Group will: 1) continue to receive usual care; 2) are eligible to receive financial incentives based on completion of recommended ADA benchmarks and achievement of goals that are founded on evidence based guidelines for diabetes; and 3) be compensated for completion of surveys.
  Interventions: Behavioral: Financial Incentives
- Control Group (No Intervention): Participants (161) in the Control Group will continue to receive usual care and be compensated for the completion of surveys only. They will not receive financial incentives.

INTERVENTIONS:
Behavioral: Financial Incentives — This intervention will examine the effects of incentives on improving adult diabetic Medicaid beneficiaries' health outcomes and reducing associated costs through healthy behavior changes in their diabetes self-management. Incentives focus on improving self-management of diabetes, compliance with ADA recommended preventive, treatment and management measures, primary biometric measures of diabetes, and eliminating barriers to a healthy lifestyle
  Arms: Financial Incentives Group

SUMMARY:
The purpose of this randomized controlled trial (RCT) study is to examine the extent that financial incentives when combined with diabetes evidence-based practices, improve self-management and biometric measures for adult diabetic Medicaid recipients with an HbA1c of ≥ 6.5 at enrollment. The study will also evaluate the cost-effectiveness of the program.

Specific Aims:

1. Evaluate whether financial incentives for completing American Diabetes Association (ADA) recommended tests, exams, health education, biometric outcome goals, and vaccinations will improve primary biometric outcomes.
2. Evaluate whether financial incentives for completing ADA recommended tests, exams, health education, biometric outcome goals, and vaccinations will improve diabetes patients' self-management as assessed by Summary of Diabetes Self-Care Activities Measure (SDSCA) and 36-Item Short Form Health Survey (SF36v2).
3. Evaluate the extent to which financial incentives for healthy behaviors reduce the cost of health care utilization.

DETAILED DESCRIPTION:
Diabetes is the seventh leading cause of death in the United States (OECD 2013). It is also known that certain populations are at greater risk for diabetes. In Hawaii, diabetes disproportionally affects Native Hawaiians and Pacific Islanders as they are three times more likely to be diagnosed with diabetes. In addition, in 2010 the U.S. Department of Health and Human Services Office of Minority Health reported that Native Hawaiians/Pacific Islanders in Hawaii were 5.7 times as likely as Caucasians living in Hawaii to die from diabetes(Office of Minority Health, 2010).

In order to address the challenges that chronic diseases impose on individuals and the health care system the Centers for Medicare & Medicaid Services (CMS) is assessing the impact of incentivizing patients to increase self-care and disease management. Previous studies have demonstrated that monetary incentives have been associated with an improvement in behavioral outcomes, most notably when the incentive is received immediately following the targeted behavior (Volpp, K.G., et.al., 2008; Mitchell, M.S., et.al., 2013). Cahill et al. (2008) showed that economic incentives were tied to smoking cessation and led to a decrease in relapse within a year. Our study seeks to build on these findings and determine whether financial incentives may provide a way to improve diabetes self-management.

Data:

Electronic data (Labs, Outcomes) - January 1st, 2013 through December 31, 2015 Electronic data (Claims) - January 1st, 2011 through December 31, 2015

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with diabetes mellitus
2. 18 years of age or older
3. Medicaid recipient
4. At recruitment has an HbA1c level of ≥ 6.5
5. At recruitment is receiving care coordination at Kaiser Permanente Hawaii

Exclusion Criteria:

1. Current pregnancy - gestational diabetes
2. End-stage Renal Disease
3. Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritabelle Fernandes, MD, Principal Investigator — University of Hawaii; Rebecca R. Ozaki, PhD, Principal Investigator — Unversity of Hawaii - Center on Disability Studies
Locations (1):
- Kaiser Permanente Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Background] Organisation for Economic Co-Operation and Development (OECD), "Health Status: Life Expectancy at Birth, in Health at a Glance 2013: available at http://www.oecd.org/els/health-systems/Health-at-a-Glance-2013.pdf.
- [Background] Office of Minority Health 2010. Diabetes Data/Statistics. Retrieved from http://minorityhealth.hhs.gov/templates/browse.aspx?lvl=3&lvlid=62
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Mitchell MS, Goodman JM, Alter DA, John LK, Oh PI, Pakosh MT, Faulkner GE. Financial incentives for exercise adherence in adults: systematic review and meta-analysis. Am J Prev Med. 2013 Nov;45(5):658-67. doi: 10.1016/j.amepre.2013.06.017. PMID 24139781
- [Background] Cahill K, Perera R. Competitions and incentives for smoking cessation. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD004307. doi: 10.1002/14651858.CD004307.pub3. PMID 18646105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited 320 eligible patients from Kaiser Permanente Hawaii. Participants were randomly assigned into the intervention or control group with 159 and 161 in each group respectively. The randomized control trial (RCT) was conducted from May 2014 to December 31, 2015 with rolling enrollment from May 2014 to January 2015.
Groups:
- Financial Incentives: Participants (159) in the Incentive Group will: 1) continue to receive usual care; 2) are eligible to receive financial incentives based on completion of recommended American Diabetes Association (ADA) benchmarks and achievement of goals that are founded on evidence based guidelines for diabetes; and 3) be compensated for completion of surveys.
  Financial Incentives: This intervention will examine the effects of incentives on improving adult diabetic Medicaid beneficiaries' health outcomes and reducing associated costs through healthy behavior changes in their diabetes self-management. Incentives focus on improving self-management of diabetes, compliance with ADA recommended preventive, treatment and management measures, primary biometric measures of diabetes, and eliminating barriers to a healthy lifestyle.
- Control: Participants (161) in the Control Group will continue to receive usual care and be compensated for the completion of surveys only. They will not receive financial incentives.
Period: Overall Study
Arm/Group | Financial Incentives | Control
Started | 159 | 161
Completed | 125 | 131
Not Completed | 34 | 30
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost Medicaid eligibility | 29 | 22
Not completed — Switched Managed Care Organization (MCO) | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Financial Incentives: Participants (159) in the Incentive Group will: 1) continue to receive usual care; 2) are eligible to receive financial incentives based on completion of recommended ADA benchmarks and achievement of goals that are founded on evidence based guidelines for diabetes; and 3) be compensated for completion of surveys.
  Financial Incentives: This intervention will examine the effects of incentives on improving adult diabetic Medicaid beneficiaries' health outcomes and reducing associated costs through healthy behavior changes in their diabetes self-management. Incentives focus on improving self-management of diabetes, compliance with ADA recommended preventive, treatment and management measures, primary biometric measures of diabetes, and eliminating barriers to a healthy lifestyle.
- Total: Total of all reporting groups
Arm/Group | Financial Incentives | Control | Total
Number analyzed (Participants) | 159 | 161 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (10.7) | 47.8 (10.0) | 48.1 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 86 | 174
  Male | 71 | 75 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 14 | 24
  Not Hispanic or Latino | 145 | 144 | 289
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 32 | 36 | 68
  Native Hawaiian or Other Pacific Islander | 54 | 48 | 102
  Black or African American | 1 | 1 | 2
  White | 27 | 22 | 49
  More than one race | 40 | 53 | 93
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 159 | 161 | 320
History of Hypertension [Count of Participants; unit: Participants] | 115 | 106 | 221
History of Heart Disease [Count of Participants; unit: Participants] | 14 | 20 | 34
History of Smoking or Tobacco Dependence [Count of Participants; unit: Participants] | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Changes in HbA1c From Baseline to the End of Intervention (December 2015)
Description: Changes in Hemoglobin A1c from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: Repeated measurements for each subject were used. The analysis was per protocol with all available observations for each subject included to estimate parameters in the mixed effects model. The mixed effects model approach can provide unbiased results when the type of missing data is missing at random, which is common for longitudinal studies.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
percentage of glycosylated hemoglobin | 0.0660 [-0.2158 to 0.3478] | -0.3440 [-0.6546 to -0.0334]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; Generalized estimating equation (GEE) modeling was used to examine the pre- and post-intervention changes between groups due to interventions in biometric indicators. The average change in scores over time for the intervention group was compared to that for the control group. The difference-in-differences values was assessed for significance at p = 0.05. Null hypothesis assumed no differences in the biometric measure from baseline to endpoint between groups; Test type: Superiority or Other; p = 0.0553, Generalized Estimating Equation Model; The analysis adjusted for the effects of age, race, gender, and baseline hypertension; Mean Difference (Final Values) = 0.4100, 95% CI 2-sided [-0.0092 to 0.8293], Standard Error of Mean 0.2139 — The estimates denote the differences between longitudinal changes within the treatment group and longitudinal changes within the control group

2. Primary Outcome: Changes in Systolic Blood Pressure From Baseline to the End of Intervention (December 2015)
Description: Changes in systolic blood pressure from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
mmHg | -1.3579 [-3.8541 to 1.1383] | 0.9337 [-1.9684 to 3.8358]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2416, Generalized Estimating Equation Model; Mean Difference (Final Values) = -2.2916, 95% CI 2-sided [-6.1274 to 1.5442], Standard Error of Mean 1.9571 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Changes in Diastolic Blood Pressure From Baseline to the End of Intervention (December 2015)
Description: Changes in diastolic blood pressure from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
mmHg | -2.1895 [-3.9359 to -0.4432] | -1.1002 [-2.8352 to 0.6347]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3881, Generalized Estimating Equation Model; The analysis adjusted for the effects of age, gender, race, and hypertension at baseline; Mean Difference (Final Values) = -1.0893, 95% CI 2-sided [-3.5632 to 1.3846], Standard Error of Mean 1.2622 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Changes in Total Cholesterol From Baseline to the End of Intervention (December 2015)
Description: Changes in total cholesterol from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
mg/dL | -3.9141 [-14.6584 to 6.8303] | 2.5709 [-13.1754 to 8.0336]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8617, Generalized Estimating Equation Model; The analysis adjusted for the effects of age, gender, race, and hypertension at baseline; Mean Difference (Final Values) = -1.3432, 95% CI 2-sided [-16.4517 to 13.7653], Standard Error of Mean 7.7086 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Changes in Triglycerides From Baseline to the End of Intervention (December 2015)
Description: Changes in triglycerides from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
mg/dL | 0.4843 [-48.524 to 49.4935] | 18.2713 [-8.7418 to 45.2845]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5333, Generalized Estimating Equation Model; The analysis adjusted for the effects of age, gender, race, and hypertension at baseline; Mean Difference (Final Values) = -17.7870, 95% CI 2-sided [-73.7478 to 38.1737], Standard Error of Mean 28.5519 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Changes in LDL From Baseline to the End of Intervention (December 2015)
Description: Changes in LDL from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
mg/dL | 0.4523 [-7.3542 to 6.4495] | 1.3620 [-8.9651 to 6.2410]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8620, Generalized Estimating Equation Model; The analysis adjusted for the effects of age, gender, race, and hypertension at baseline; Mean Difference (Final Values) = 0.9097, 95% CI 2-sided [-9.3509 to 11.1702], Standard Error of Mean 5.2351 — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Changes in HDL From Baseline to the End of Intervention (December 2015)
Description: Changes in HDL from baseline to end of study. Change = (End of Intervention score - Baseline score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
mg/dL | 0.6705 [-0.7934 to 2.1344] | -0.0472 [-1.4807 to 1.3863]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4915, Generalized Estimating Equation Model; The analysis adjusted for the effects of age, gender, race, and hypertension at baseline; Mean Difference (Final Values) = 0.7177, 95% CI 2-sided [-1.3272 to 2.7626], Standard Error of Mean 1.0433 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Changes in Health Utilization Cost Before and During Intervention - Amount Paid by Service Providers
Description: Changes of total cost expenditures including emergency room use and hospitalizations in the intervention and control groups before and during intervention.
Time Frame: Before intervention (3 years prior to baseline) and during intervention (2 years from baseline to end of intervention)
Measure: Mean (Standard Error); unit: dollars/day
Groups:
- Financial Incentives: Participants (159) in the Incentive Group will: 1) continue to receive usual care; 2) are eligible to receive a maximum of $320 financial incentives annually based on completion of recommended ADA benchmarks and achievement of goals that are founded on evidence based guidelines for diabetes; and 3) be compensated for completion of surveys.
  Financial Incentives: This intervention will examine the effects of incentives on improving adult diabetic Medicaid beneficiaries' health outcomes and reducing associated costs through healthy behavior changes in their diabetes self-management. Incentives focus on improving self-management of diabetes, compliance with ADA recommended preventive, treatment and management measures, primary biometric measures of diabetes, and eliminating barriers to a healthy lifestyle.
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 159 | 161
dollars/day | -0.185 (0.674) | -0.203 (0.484)
Statistical Analysis 1: Comparison: Financial Incentives vs Control; A standard diffs-in-diffs model was utilized to estimate the causal effect of the intervention on medical costs per patient/day. The average change in cost over time for the intervention group was compared to that for the control group. The difference-in-differences values was assessed for significance at p = 0.05. Null hypothesis assumed no difference in the cost per patient per day from baseline to endpoint between groups; Test type: Superiority or Other; p > 0.05, standard diffs-in-diffs model

9. Secondary Outcome: Change From Baseline to End of Intervention (December 2015) in General Diet Subscale of The Summary of Diabetes Self-Care Activities (SDSCA) Measure
Description: SDSCA is a validated, self-reported measure assessing the average # of days the recommended diabetes self-care activities are performed over the past 7 days in the areas of general diet, specific diet, exercise, blood-glucose testing, and foot care at baseline, mid, and end of intervention. Possible scores range from 0 to 7 days. Change = (End of Intervention Score - Baseline Score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: Repeated measurements for each subject were used. The analysis was per protocol with all available observations for each subject included to estimate parameters in the mixed effects model; this provides unbiased results when missing data is random. Not all participants submitted surveys at each data point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 147 | 131
units on a scale | 0.7796 [0.3492 to 1.2099] | 0.1393 [-0.3028 to 0.5814]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; The average change in scores over time for the intervention group was compared to that for the control group. The difference in these average changes is referred to as the difference-in-differences values which was assessed for significance at p = 0.05. Null hypothesis assumed no difference in the General Diet subscale from baseline to endpoint between groups. Generalized estimating equation modeling was used to examine changes in SDSCA between groups at different time points; Test type: Superiority or Other; p = 0.0420, Generalized Estimating Equation Model; Mean Difference (Final Values) = 0.6403, 95% CI 2-sided [0.0233 to 1.2572], Standard Error of Mean 0.3148 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline to End of Intervention (December 2015) in Physical Component Summary Measure of the Short Form (SF-36v2) Health Survey
Description: The SF-36v2 is validated, self reported short-form health survey used to assess changes over time in the well-being of participants. It consists of 2 component summary measures that further summarize 8 health domain scales. The Physical Component Summary (PCS) measure is derived from domain scales of Physical Functioning (10 items), Role-Physical (4 items), Bodily Pain (2 items), and General Health (5 items). Scores of component summary measures and health domain scales range from 0 to 100 with higher scores indicating better outcomes. Norm-based scoring was used so that scores for each health domain scale and component summary measure have a mean of 50 and standard deviation of 10 based on the 2009 U.S. general population. The SF-36v2 was used to assess participants' health and wellbeing at baseline, mid, and endpoint of intervention. Change = (Midpoint Score - Baseline Score)
Time Frame: Baseline to end of intervention - 12 months minimum to 19 months maximum due to rolling enrollment
Population: Repeated measurements for each subject were used. The analysis was per protocol with all available observations for each subject included to estimate parameters in the mixed effects model; this provides unbiased results when the type of missing data is random. Not all participants submitted surveys at each data point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 145 | 132
units on a scale | 0.5162 [-0.8996 to 1.9319] | -1.6027 [-3.0495 to -0.1558]
Statistical Analysis 1: Comparison: Financial Incentives vs Control; The average change in scores over time for the intervention group was compared to that of the control group. The difference in the average changes is referred to as the difference-in-differences values which was assessed for significance at p=0.05. Null assumed no group difference in the Physical Component Summary measure of SF-36v2 from baseline to midpoint. Generalized estimating equation (GEE) modeling was used to examine changes in health measures between groups at different time points; Test type: Superiority or Other; p = .0399, Generalized Estimating Equation Model; The effect of age and gender is adjusted in the GEE model; Mean Difference (Final Values) = 2.1188, 95% CI 2-sided [0.0981 to 4.1395], Standard Error of Mean 1.0310 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year 7 months
Description: The consent form detailed that participants were at no more risk than that related to standard of care. Should an adverse event have occurred due to standard of care, service providers were responsible and did not communicate any adverse events. Incentives through HI-PRAISE were based on ADA standards of care and did not increase risk. No Adverse Events were reported.
Arm/Group | Financial Incentives | Control
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/161
Other Adverse Events (participants affected / at risk) | 0/159 | 0/161

LIMITATIONS AND CAVEATS:
Loss of Medicaid status led to reduced # of data points analyzed. Unequally spaced intervention period across subjects increased the variability of outcomes. Usual care setting with providers ordering lab tests led to high # of missing test results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days